CLINICAL TRIAL: NCT02992067
Title: CK19 Combined With Contrast-enhanced Ultrasound: a Prediction System on Axillary Lymph Node Metastasis in Breast Cancer
Acronym: CK-CEUS
Status: Completed | Type: Observational
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, YU Xingfei, Breast Tumor Surgery (Department 104), Zhejiang Cancer Hospital
Other Study IDs: ZJCH-CK19A
Record Dates: First submitted 2016-12-09; First posted 2016-12-14 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Lymph Node; Breastcancer
Keywords: lymph node metastasis; breast cancer; CK19; contrast-enhanced ultrasonography
MeSH Terms: conditions — Lymphatic Metastasis; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Operable breast cancer: clinical stage: cTis, cI, cII, cT3N1M0

SUMMARY:
To establish a predicting system on axillary lymph node metastasis based on peripheral blood CK19mRNA and contrast-enhanced ultrasound.

DETAILED DESCRIPTION:
The feasibility and predictive accuracy of peripheral blood CK19mRNA and contrast-enhanced ultrasound of axillary lymph nodes metastasis in breast cancer were verified by the data of specimen bank; to establish the evaluation system of predicting the lymph node status based on CK19 and CEUS, validate the sensitivity, specificity, negative predictive value, positive predictive value and ROC curve of the system model and use Youden index, negative likelihood ratio, positive likelihood ratio to evaluate the diagnostic efficiency.

ELIGIBILITY:
Inclusion Criteria:

1. female, age 18~70 years old
2. the test group should be in accordance with the pathological diagnosis of breast cancer, the clinical stage of breast cancer (stage cTis, cI, cII and cT3N1M0), the initial treatment to receive surgical treatment. Complete preoperative clinical diagnosis data, including the ipsilateral axillary lymph node CEUS data and peripheral blood sample; The negative-control group should comply with the pathological diagnosis, breast adenosis, fibrocystic lesions, breast cysts and other benign lesions, with complete preoperative clinical data, also including ipsilateral axillary lymph node CEUS data and peripheral blood sample

Exclusion criteria:

1. metastatic breast cancer, inflammatory breast disease, surgery without lymph node staging
2. pregnancy or lactation
3. patients with hematopoietic system disease or cancer, autoimmune diseases
4. preservation of substandard peripheral blood samples.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Operable breast cancer patients (clinical stage: cTis, cI, cII, cT3N1M0)
Sampling Method: Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xingfei Yu, M.D., Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qiao E, Yu X, Zhou L, Wang C, Yang C, Yu Y, Chen D, Huang J, Yang H. A Prospective Validation Cohort Study of a Prediction Model on Non-sentinel Lymph Node Involvement in Early Breast Cancer. Ann Surg Oncol. 2020 May;27(5):1653-1658. doi: 10.1245/s10434-019-07980-x. Epub 2019 Oct 28. PMID 31659631

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Operable Breast Cancer
Started | 359
Completed | 359
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Operable Breast Cancer
Number analyzed (Participants) | 359
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.88 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 359
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 359
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 359
Lymph node involvement [Count of Participants; unit: Participants] | 359

OUTCOME MEASURES:

1. Primary Outcome: The Accuracy of CK19 Combined With Contrast-enhanced Ultrasound (CEUS) Predicting Value on Involved Lymph Node
Description: The accuracy means the conformity of predicting results and the pathological result in lymph node involvement and also the false negative rate of sentinel lymph node (SLN) and non-SLN (nSLN) using prediction model by CK19 combined with CEUS examination
Time Frame: 1 year
Measure: Number; unit: proportion of false negative lymphnodes
Arm/Group | Operable Breast Cancer
Number analyzed (Participants) | 359
proportion of false negative lymphnodes | 0.0896

ADVERSE EVENTS:
Time Frame: 1year
Arm/Group | Operable Breast Cancer
All-Cause Mortality (participants affected / at risk) | 0/359
Serious Adverse Events (participants affected / at risk) | 0/359
Other Adverse Events (participants affected / at risk) | 0/359

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT02992067/Prot_SAP_000.pdf